CLINICAL TRIAL: NCT05366972
Title: Evaluation of Morphological Features of Thoracolumbar Fascia by Ultrasonography in Patients With Low Back Pain
Brief Title: Measuring the Morphological Characteristics of Thoracolumbar Fascia in Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Assoc.Phd.M.D, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2020/06-24
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients diagnosed with low back pain (Active Comparator): Measurements of the back muscles and thoracolumbar fascia will be made by ultrasonography.
  Interventions: Device: Ultrasonographic measurements
- Healthy volunteers (Active Comparator): Measurements of the back muscles and thoracolumbar fascia will be made by ultrasonography.
  Interventions: Device: Ultrasonographic measurements

INTERVENTIONS:
Device: Ultrasonographic measurements — Posterior layers of the thoracolumbar fascia ,middle layers of the thoracolumbar fascia thickness and Lumbar interfacial triangle thickness
  CSA (cross-sectional area) measurements of erector spinae muscles, quadratus lumborum muscles and the latissimus dorsi muscles

SUMMARY:
Recently, it has been reported that the thoracolumbar fascia may play a role in the pathophysiology of chronic low back pain.There is still no standard method for imaging and analyzing the thoracolumbar fascia.The aim of this study is to advance the understanding of the role of the thoracolumbar fascia in chronic low back pain as well as to advance the analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Patients with low back pain for more than 6 months
* Healthy volunteers

Exclusion Criteria:

* Previous low back or back surgery
* Uncontrolled Diabetes Mellitus
* Mental retardation
* Metabolic disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-10 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
fascia thickness | 20 minutes
  The posterior, middle layer thoracolumbar fascia thickness and Lumbar interface triangle thickness were determined by ultrasonography.

SECONDARY OUTCOMES:
CSA | 20 minute
  CSA (Sectional Area) measurements of erector spina ,quadratus lumborum and latissimus dorsi muscles by ultrasonography
VAS | 20 minutes
  visual analog scale (VAS) :for pain. 0: no pain at all, 10: worst pain imaginable
ODİ | 30 minutes
  Oswestry Disability Index Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.(1)

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Metin Ökmen, Assoc. PhD., Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

REFERENCES:
- [Result] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683